CLINICAL TRIAL: NCT02897700
Title: A Phase I Multi-Center Study to Evaluate the Safety, Tolerability, and Efficacy of Chemotherapeutic Regiments in Surgical Patients With Infiltrating Ductal Carcinoma of Breast
Brief Title: A Randomized Trial of Chemotherapy in Surgical Patients With Infiltrating Ductal Carcinoma of Breast
Acronym: COC-IDCB
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai 10th People's Hospital (Other); China-Japan Union Hospital, Jilin University (Other); Ganzhou City People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Sun, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCA-81472709
Record Dates: First submitted 2016-08-25; First posted 2016-09-13 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Safety; Tolerability; Efficacy
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Epirubicin; Fluorouracil; Methotrexate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mono-chemotherapy (Experimental): A mono-chemotherapy (a single chemotherapeutic agent out of cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (or CDEFM) was performed 30~60 days prior to surgery for patients who had no history of receiving either local or systemic cancer-associated chemotherapy.
  Interventions: cyclophosphamide, doxorubicin, epirubicin, fluorouracil or methotrexate.
  Interventions: Drug: Single agent of cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate
- Combined chemotherapy (Experimental): Combined chemotherapy (random combination of two breast cancer chemotherapeutic agents including cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate, or CDEFM) was performed 30~60 days prior to surgery for patients who had no history of receiving either local or systemic chemotherapy for cancer.
  Interventions: cyclophosphamide, doxorubicin, epirubicin, fluorouracil or methotrexate.
  Interventions: Drug: cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (CDEFM)
- Placebo treatment (Placebo Comparator): No chemotherapeutic regimes using any cytotoxic agent was done for patients who have infiltrating ductal carcinoma of breast. Placebo was used instead.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Single agent of cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate — Procedure: Routine chemotherapeutic regimens using one out of cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (CDEFM) as single agent was performed 30~60 days before surgery：cyclophosphamide 100mg/M2, doxorubicin 60mg/M2, epirubicin 100mg/M2, fluorouracil 500mg/M2, or methotrexate 50mg/M2.The agent was given on a regular route of IV administration on the 1st and 8th day of each cycle, 28 days per cycle, totally 6 cycles. Subsequently, there was a 30-day interval between the last cycle and radical surgery.
  Arms: Mono-chemotherapy
Drug: cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (CDEFM) — Procedure: Routine chemotherapeutic regimens using two agents from cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (CDEFM) as combinatorial treatment was performed 30~60 days before surgery：cyclophosphamide 100mg/M2, doxorubicin 60mg/M2, epirubicin 100mg/M2, fluorouracil 500mg/M2, or methotrexate 50mg/M2.The agents were given on a regular route of IV administration on the 1st and 8th day of each cycle, 28 days per cycle, totally 6 cycles. Subsequently, there was a 30-day interval between the last cycle and radical surgery.
  Arms: Combined chemotherapy
Drug: Placebo — Procedure: Routine placebo standardized in clinical oncology was provided to patients to replace any chemotherapeutic agent.
  Arms: Placebo treatment

SUMMARY:
The overarching purpose of this study is to determine if the mainstay chemotherapeutic regimens represented by several genotoxic agents including but not limited to Cyclophosphamide, Doxorubicin, Epirubicin, Fluorouracil and Methotrexate (CDEFM), in the format of either a single agent or combinations are safe, tolerable, and effective in the treatment of patients with infiltrating ductal carcinoma of breast.

DETAILED DESCRIPTION:
Infiltrating ductal carcinoma (IDC) of breast, or sometimes called invasive ductal carcinoma of breast, is the most common type of breast malignancy. About 80% of all breast cancers are IDCs.

Once found, IDC usually has already broken through the wall of the milk duct and begun to invade the tissues of the breast. Over time, IDC can spread to the lymph nodes and possibly to other areas of the body with high frequency.

According to the statistics of American Cancer Society, more than 180,000 women in the United States are diagnosed with IDC each year. Although IDC can affect women at any age, it is more common as they grow older. Further, approximately two-thirds of women are 55 or older when they are diagnosed with such this symptom.

The treatments for invasive ductal carcinoma fall into two broad categories. First, local treatments for IDC, including surgery and radiation, which treat the primary tumor and surrounding areas such as the chest and lymph nodes. Second, systemic treatments for IDC, including chemotherapy, hormone therapy and targeted therapy, which are supposed to deliver cytotoxicity throughout the body to eliminate any cancer cells that have left the primary site and to help minimize the risk of recurrent disease.

PURPOSE: This randomized phase I trial is to determine the safety, tolerability and efficacy of single or concurrent administration of cyclophosphamide, doxorubicin, epirubicin, fluorouracil and methotrexate (CDEFM) to women undergoing surgery for infiltrating ductal carcinoma in situ breast cancer.

RATIONALE: This is a randomized, controlled, open-labeled and multicenter, pilot study. Patients are randomized to 1 of 2 treatment arms (arms A or B). Patients accrued as control participants are assigned to arm C. to implement the study, the investigators will collect surgical samples of the primary tumor and periphery blood from breast cancer patients to assess the effects of chemotherapeutic regimens and correlation with post-therapy survival in the patient cohorts. Besides the five-year disease-free survival, overall survival and five-year metastasis-free survival post treatment, the investigators also analyze and evaluate the anticancer agent-induced tumor stroma damage extent, which may provide further evidence to confirm the treatment efficacy and appraise the potential influence of a damaged tumor microenvironment on disease progression or regression in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with histologically proven infiltrating ductal carcinoma of breast
* no severe major organ dysfunction
* Patients must have adequate hematopoietic function as evidenced by:

white blood cells (WBC) ≥ 3,000/μl absolute neutrophil count (ANC) ≥ 1,500/μl Platelet count ≥ 100,000/μl hemoglobin (HGB) ≥ 10 g/dl and not transfusion dependent

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 10% above upper limit of normal
* Individuals of child-bearing potential must have a negative serum or urine pregnancy test within 72 hours of Cycle 1 Day 1.
* World Health Organization (WHO) performance status of 0 or 1
* No prior or concurrent cancer-associated chemotherapy, no initiation of new hormonal therapy
* Hormone receptor (estrogen receptor (ER), progesterone receptor (PR), epidermal growth factor receptor 2 (Her2)) status not specified
* Menopausal status not specified
* Patients or their legal representatives must be willing and able to provide written informed consent
* A Clinical Stage ≥ I subtype A (IA) (T1a, N0, M0) of Beast Cancer but without diagnosed distant metastasis (according to the 1997 revision of the International Union Against Cancer-PrimaryTumor, Regional Nodes and Metastasis (TNM) staging system) as determined by a preoperative evaluation that included a chest computed tomography (CT) scan and/or X-ray mammography.

Exclusion Criteria:

* Age < 18
* Severe major organ dysfunction
* WHO performance status of >1
* Prior cancer chemotherapy
* Stage IV
* Patients with symptomatic central nervous system (CNS) metastases from breast cancer
* Patients with a history of another invasive malignancy within the last 3 years
* History of loss of consciousness or transient ischemic attack within 12 months before study treatment initiation.
* Patients who have known active HIV, Hepatitis B, or Hepatitis C infections.
* Patients with any other condition which in the opinion of the investigator would preclude participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 months
  The case of emergent events caused by treatment is measured by counting the blood cell number and detecting liver and kidney functions. Total blood cell number, alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT) and lactate dehydrogenase (LDH) > 20% above upper limit of normal, is considered as not safe.
  Tolerability is measured by monitoring the first occurrence of grade 4 hematologic or grade 3-4 non hematologic toxicity as defined by the National Cancer Institute (NCI)-Common Toxicity Criteria (CTC) (NCI-CTC version 4; or CTCAE v4.0) and/or disruption of chemotherapy because of inacceptable toxicity.
  Chemotherapeutic efficacy is measured by the remaining tumor size after computed tomography (CT) scanning and comparing it with the original primary tumor size 2-3 weeks after last cycle of chemotherapy. The ratio of post-treatment tumor size to pre-treatment tumor size < 50% is considered as effective. Otherwise not.

SECONDARY OUTCOMES:
Circulating concentrations of tumor microenvironment-specific soluble factors | 6 months
  Influence of the cytotoxicity of chemotherapeutic regimens on the primary tumor microenvironment is systemically measured for each patient. The circulating amounts per volume of a group of literature-reported soluble factors including interleukin (IL)-6, IL-8, granulocyte macrophage colony stimulating factor (GM-CSF), Wnt family member 16B (WNT16B) and serine peptidase inhibitor Kazal type 1 (SPINK1) are measured in the peripheral blood 2-3 weeks post treatments to assess the influence of chemotherapies. Concentration of either IL-6 > 50 ng/ml, IL-8 > 80 ng/ml, GM-CSF > 20 ng/ml, WNT16B > 100 ng/ml or SPINK1 > 60 ng/ml, is considered that the primary tumor has an activated microenvironment. The measurement continues for two more times, including one performed at 2 months and the other performed as 6 months after completion of chemotherapeutic regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (3):
- China (3):
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi
  - China-Japan Union Hospital, Jilin University, Changchun, Jilin
  - Shanghai 10th People's Hospital, Tongji University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Output data from this clinical study will be be made available to the public appropriately upon complete of the primary investigation, according to the original plan.